CLINICAL TRIAL: NCT07391813
Title: A Phase 1b/2, Open-Label, Multi-center Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of SNB-101, in Extensive Stage Small Cell Lung Cancer.
Brief Title: SNB-101 for Treatment of Extensive Stage Small Cell Lung Cancer
Acronym: SNB-101-101
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SN BioScience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SNB-101-101*
Record Dates: First submitted 2026-01-17; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Patient is Not Suitable for Complete Surgical Resection With a Cytologically or Histologically Confirmed Small Cell Lung Cancer(SCLC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Participants receive SNB-101 administered intravenously according to the study protocol.
  Interventions: Drug: SNB-101

INTERVENTIONS:
Drug: SNB-101 — SNB-101 is a nanoparticle formulation of SN-38 administered intravenously. Subject enrolled for each dose level cohort of 50/80 mg/m2, 60/96 mg/m² and 70/112 mg/m2 will be administered intravenously over 90 minutes at Day 1 and Day 15 of each cycle

SUMMARY:
The purpose of the Phase 1 research is to test the safety, tolerability, maximum tolerated dose, and pharmacokinetics (PK- the study of how a medicine moves through subject body. It looks at how the drug is absorbed, travels in your blood, reaches different parts of subject body, and is eventually broken down and removed) of the SNB-101.The Phase 2 is to determine the optimal dose (amount of medicine that works best to treat a condition while causing the fewest side effects) of SNB-101 for further research and to collect a further information on PK, safety and tolerability.

Once subject has completed assessments during screening and if subject is found eligible to participate in the study, study drug will be given by intravenous infusion on day 1 and day 15 of each cycle treatment.

Throughout the treatment period, the study doctor will monitor subject for any changes to subject health. While subject is taking the study drug, we will ask subject the following:

* How subject are feeling.
* If subject has experienced any side effects.
* If subject is taking other medications or if there are changes to the medications subject was taking before.

The study drug will be taken over multiple cycles. A cycle is the time between the start of 1 round of treatment until the start of the next round. In this study, each treatment cycle is of 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients over 18 years of age.
2. Male or fertile female patients who have agreed to comply with effective contraceptive methods as required by this protocol and the specified contraceptive period.
3. Participants must have a cytologically or histologically confirmed small cell lung cancer which is locally advanced or metastatic and has progressed on or after standard therapy for advanced disease containing platinum-based therapy plus etoposide with or without atezolizumab or durvalumab immunotherapy and is not suitable for complete surgical resection.
4. Have measurable or evaluable disease consistent with RECIST (Response Evaluation Criteria in Solid Tumors) version 1.1
5. With life expectancy more than 12 weeks
6. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
7. Have adequate hematological, renal, and liver function as defined by the following (lab test can be repeated during screening):
8. Have recovered to grade 1 or better to (CTCAE version 5.0) from any reversible side effects of previous treatments. Note: Grade 2 alopecia and Grade 2 sensory neuropathy are not exclusionary.
9. No major surgery, no antineoplastic or experimental therapy, and no direct radiation therapy to a hematopoietic site within 4 weeks prior to baseline, and no biologic drugs, nitrosoureas or mitomycin C administered within 6 weeks prior to baseline.
10. Fully informed regarding the investigational nature of the study protocol and is capable of signing an Institutional Review Board/Ethics Committee-approved informed consent form.

Exclusion Criteria:

1. Patients in whom the homozygous variant alleles UGT1A1*28 or UGT1A1*6 are confirmed through UGT1A1 genotype testing at screening (or through previously conducted testing), or patients with heterozygous variant alleles UGT1A1*6/*28. (For Phase 1 only)
2. Female patients who are pregnant, lactating (breast feeding) or planning a pregnancy during the course of study.
3. Known or suspected intolerance or hypersensitivity to the main ingredient or any of the excipients of SNB-101.
4. Patients deemed unsuitable or ineligible for participation in this clinical trial as judged by the Principal Investigator.

   Medical History or Current Pathological Conditions and Diseases
5. Known uncontrolled symptomatic heart failure.
6. History of alcohol abuse or other substance abuse within 1 year prior to screening.
7. Have intestinal palsy or bowel obstruction.
8. Have chronic inflammatory bowel disease.
9. Are on dialysis.
10. Patients with any evidence of current ILD or pneumonitis or a prior history of interstitial lung disease (ILD) or non-infectious pneumonitis requiring high-dose glucocorticoids.
11. Patients with clinically significant congestive heart failure that is uncontrolled.
12. Have multiple ascites or pleural effusion.
13. Have hematologic malignancy (including lymphoma).
14. Have severe infections or other uncontrolled active infections that require the administration of antibiotics, antivirals, or other anti-infective agents that may affect safety or efficacy assessments during the clinical study, as determined by the investigator.
15. When the QTc interval exceeds 480 msec* (same standard for both men and women). * Fridericia's QT correction formula
16. Positive for Human Immunodeficiency Virus (HIV).
17. Patients with known active hepatitis B (e.g., HBsAg response positive and HBV DNA detected) or hepatitis C (e.g., anti-HCV positive and HCV RNA [qualitatively]) detected).
18. Central nervous system or brain metastases with clinically significant symptoms requiring systemic corticosteroids at least 2 weeks prior to baseline. (however, participants who have completed treatment and recovered from the acute phase of radiation therapy or surgery may participate in this study.).

    Patients Who Have Received, are Receiving, or Cannot Discontinue the Following Medications or Therapies.
19. Have received another investigational drug within the last 4 weeks prior to screening.
20. If additional anticancer therapy* other than the investigational drug is required during the clinical trial participation period. (However, localized radiation therapy for palliation purposes, such as for bone pain, bronchial obstruction, or skin lesions, is allowed).
21. Surgery, radiation (chemotherapy), chemotherapy, targeted therapy (small molecule drugs, monoclonal antibodies), immunotherapy (biological agents), or hormone therapy, etc.
22. If strong CYP3A4 inducer was administered within 2 weeks before baseline : (Phenytoin, carbamazepine, rifamycin (rifampicin, rifabutin, rifapentine), phenobarbital, etc., Preparations containing St. John's wort.
23. Have received a strong CYP3A4 and/or UGT1A1 inhibitor (azole antifungal agents [ketoconazole, fluconazole, itraconazole, miconazole, voriconazole, etc.], macrolide antibiotics [erythromycin, clarithromycin, etc.], antiretroviral agents [atazanavir, ritonavir, indinavir, lopinavir, nelfinavir, saquinavir, telaprevir], sorafenib, diltiazem hydrochloride, nefazodone, gemfibrozil, nifedipine, etc., or grapefruit juice) within 1 week prior to baseline
24. Will require administration of neuromuscular blockers, peripheral muscle relaxants, etc. during the study : Non-depolarizing neuromuscular blockers (such as succinylcholine) and depolarizing neuromuscular blockers (such as rocuronium)
25. Will require lapatinib during the study.
26. When administration of live herbal medicine detoxified vaccine is required during the clinical trial participation period: Yellow fever vaccine, etc.
27. Are taking a drug during the study that in the judgment of the investigator will have a significant effect on liver metabolism or kidney excretion. However, taking such a drug is permitted if (a) it was taken more than 4 weeks prior to baseline.
28. If the participant is deemed to be taking medications (including over-the-counter drugs, herbs, or homeopathic remedies) that significantly affect the action, metabolism, and excretion of the IP, as well as its efficacy and safety of the IP, as determined by the investigator. (However, if the participant has been taking the same dose of medication for at least 1 week prior to baseline [excluding drugs taken daily; if taken regularly or periodically, it is included], they are exempt).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) according to CTCAE version 5.0 in Phase 1 | Dose limiting toxicities will be evaluated during the first treatment cycle (28 days)
  Nature and frequency of dose-limiting toxicities (DLTs) associated with SNB-101 administration
Treatment discontinuation/dose reduction due to Adverse Events (AEs) in Phase 1 | Day 1 through study completion, an average of 2 years
  Number of participants who permanently discontinue or dose reduction of SNB-101 because of adverse events.
Number of Adverse Events (AE) that occurs in Phase 1Number of Adverse Events (AE) that occurs in Phase 1 | Adverse events will be recorded from informed consent through 28 days (±7 days) after the last dose of study drug
  All AEs will be graded according to CTCAE version 5.0 Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe or medically significant but not immediately life-threatening, Grade 4: Life-threatening consequences Grade 5: Death related to AE
Laboratory Parameters in Phase 1 | For hematology, clinical chemistry and coagulation: at Screening; at Days 1, 8, 15, and 22 of Cycle 1; at Days 1 and 15 of each subsequent treatment cycle (each cycle is 28 days); and at End of Treatment (EOT) For urinanalysis: at screening, day 1 of cy
  Incidence of clinically significant clinical laboratory abnormalities (hematology, clinical chemistry, coagulation, and urinalysis)
Vital Signs in Phase 1 | Baseline through study completion, an average of 2 years
  Incidence of clinically significant vital signs abnormalities, including blood pressure, heart rate, respiratory rate, and body temperature.
ECG Parameters in Phase 1 | On Day 1 of cycle 1, cycle 2, cycle 3 and cycle 4. (Each cycle is 28 days)
  Incidence of clinically significant 12-lead ECG abnormalities, assessed from triplicate ECG recordings, including QT/QTc interval
Chest X-ray (CXR) Abnormalities in Phase 1 | Baseline (Screening) through study completion, an average of 2 years
  Incidence of clinically significant chest X-ray abnormalities.
Optimized Dose of SNB-101 in Phase 2 | Day 1 through study completion, an average of 2 years
  Determination of optimized dose based on totality of data including safety/tolerability, dose intensity, need for modifications, and preliminary efficacy from two dose levels.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) in Phase 1 and 2 | At every 2 cycles (each cycle is 28 days) from baseline (Cycle 1 Day 1) until disease progression or initiation of subsequent chemotherapy (up to 2 years).
  Objective Response Rate defined as the proportion of participants with Complete Response (CR) or Partial Response (PR) per RECIST v1.1, as assessed by the Investigator.
Duration of Response (DOR) in Phase 1 and 2Duration of Response (DOR) in Phase 1 and 2 | At every 2 cycles (each cycle is 28 days) from baseline (cycle 1 day 1) until disease progression or initiation of subsequent chemotherapy (up to 2 years).
  Duration of Response defined as the time from first documented response (CR or PR) to first evidence of disease progression or death from any cause, per RECIST v1.1, as assessed by the Investigator.
Progression-Free Survival (PFS) in Phase 1 and 2 | At every 2 cycles (each cycle is 28 days) from baseline (Cycle 1 Day 1) until disease progression or initiation of subsequent chemotherapy (up to 2 years).
  Progression-Free Survival defined as the time from first dose (C1D1) to first documented disease progression or death from any cause, per RECIST v1.1, as assessed by the Investigator.
Overall Survival (OS) in Phase 1 and 2 | Upto 2 years
  Overall Survival defined as the time from first dose (C1D1) to death.
Disease Control Rate (DCR) Phase 1 | At every 2 cycles (each cycle is 28 days) from baseline (Cycle 1 Day 1) until disease progression or initiation of subsequent chemotherapy (up to 2 years).
  Disease Control Rate defined as the proportion of participants with best overall response of CR, PR, or Stable Disease (SD) per RECIST v1.1, as assessed by the Investigator.
Overall Survival Rate at 12 Months in Phase 2 | 12 months
  Proportion of participants alive at 12 months from first infusion.
Maximum plasma concentration [Cmax] in Phase 1 and 2 | Up to 168 hours post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (each cycle is 28 days); and up to 24 hours post-dose on Cycle 2 Day 1 and Cycle 4 Day 1 (sparse sampling; each cycle is 28 days).
  Pharmacokinetic profile of SNB-101 (Irinotecan, SN-38 (encapsulated and free), SN-38G) measured by Cmax
Time to maximum plasma concentration [tmax] in Phase 1 and 2 | Up to 168 hours post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (each cycle is 28 days); and up to 24 hours post-dose on Cycle 2 Day 1 and Cycle 4 Day 1 (sparse sampling; each cycle is 28 days).
  Pharmacokinetic profile of SNB-101 (Irinotecan, SN-38 (encapsulated and free), SN-38G) measured by tmax
Last Measurable Plasma Concentration (Clast) in Phase 1 and 2 | Up to 168 hours post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (each cycle is 28 days); and up to 24 hours post-dose on Cycle 2 Day 1 and Cycle 4 Day 1 (sparse sampling; each cycle is 28 days).
  Pharmacokinetic profile of SNB-101 (Irinotecan, SN-38 (encapsulated and free), SN-38G) measured by Clast
Time of Last Measurable Concentration (Tlast) in Phase 1 and 2 | Up to 168 hours post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (each cycle is 28 days); and up to 24 hours post-dose on Cycle 2 Day 1 and Cycle 4 Day 1 (sparse sampling; each cycle is 28 days).
  Pharmacokinetic profile of SNB-101 (Irinotecan, SN-38 (encapsulated and free), SN-38G) measured by Tlast
Area under the concentration-time curve from zero to a definite time [AUC(0-t)] in Phase 1 and 2 | Up to 168 hours post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (each cycle is 28 days); and up to 24 hours post-dose on Cycle 2 Day 1 and Cycle 4 Day 1 (sparse sampling; each cycle is 28 days).
  Pharmacokinetic profile of SNB-101 (Irinotecan, SN-38 (encapsulated and free), SN-38G) measured by AUC(0-t)
Area under the concentration-time curve from zero to an infinite time [AUC(0-inf)] in Phase 1 and 2 | Up to 168 hours post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (each cycle is 28 days); and up to 24 hours post-dose on Cycle 2 Day 1 and Cycle 4 Day 1 (sparse sampling; each cycle is 28 days).
  Pharmacokinetic profile of SNB-101 (Irinotecan, SN-38 (encapsulated and free), SN-38G) measured by AUC(0-inf)
Elimination half-life [t1/2] in Phase 1 and 2 | Up to 168 hours post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (each cycle is 28 days); and up to 24 hours post-dose on Cycle 2 Day 1 and Cycle 4 Day 1 (sparse sampling; each cycle is 28 days).
  Pharmacokinetic profile of SNB-101 (Irinotecan, SN-38 (encapsulated and free), SN-38G) measured by t1/2
Clearance (CL/F) in Phase 1 and 2 | Up to 168 hours post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (each cycle is 28 days); and up to 24 hours post-dose on Cycle 2 Day 1 and Cycle 4 Day 1 (sparse sampling; each cycle is 28 days).
  Pharmacokinetic profile of SNB-101 (Irinotecan, SN-38 (encapsulated and free), SN-38G) measured by CL/F
Elimination Rate Constant (Ke) in Phase 1 and 2 | Up to 168 hours post-dose on Cycle 1 Day 1 and Cycle 3 Day 1 (each cycle is 28 days); and up to 24 hours post-dose on Cycle 2 Day 1 and Cycle 4 Day 1 (sparse sampling; each cycle is 28 days).
  Pharmacokinetic profile of SNB-101 (Irinotecan, SN-38 (encapsulated and free), SN-38G) measured by Ke
Inter-individual Variability in Clearance (CL/F) in Phase 2 | Day 1 through study completion, an average of 2 years
  Inter-individual variability in apparent clearance (CL/F) across participants estimated using population pharmacokinetic modeling.
Population Clearance (CL/F) of SNB-101 in Phase 2 | Day 1 through study completion, an average of 2 years
  Apparent population clearance (CL/F) of irinotecan, SN-38 (encapsulated and free), and SN-38G estimated using population pharmacokinetic modeling based on sparse and intensive plasma concentration sampling.
Population Volume of Distribution (V/F) of SNB-101 in Phase 2 | Day 1 through study completion, an average of 2 years
  Apparent population volume of distribution (V/F) of irinotecan, SN-38 (encapsulated and free), and SN-38G estimated using population pharmacokinetic modeling.
Exposure-Response Relationship in Phase 2: Correlation Between SN-38 Exposure (AUC0-t) and Objective Response Rate (ORR) | Up to 24 months tumour assessments every 2 cycles [every 8 weeks ±7 days]; each cycle is 28 days).
  Correlation between SN-38 systemic exposure measured by AUC0-t and ORR (CR/PR) per RECIST v1.1, assessed by Investigator.
Exposure-Response Relationship in Phase 2: Correlation Between SN-38 Exposure (AUC0-t) and Incidence of TEAEs in Phase 2 | Day 1 through study completion, an average of 2 years
  Correlation between systemic exposure to SN-38 measured by area under the plasma concentration-time curve from 0 to last measurable concentration (AUC0-t) and incidence of treatment-emergent adverse events (TEAEs) (TEAEs graded per NCI CTCAE v5.0).
Treatment modification/discontinuation/dose reduction due to intolerable side effects in Phase 2 | Adverse events will be recorded from informed consent through 28 days (±7 days) after the last dose of study drug
  Number of participants who modify, discontinue or reduction of SNB-101 because of adverse events.
Number of Adverse Events (AE) that occurs in Phase 2 | Adverse events will be recorded from informed consent through 28 days (±7 days) after the last dose of study drug
  All AEs will be graded according to CTCAE version 5.0 Grade 1: Mild, Grade 2: Moderate, Grade 3: Severe or medically significant but not immediately life-threatening, Grade 4: Life-threatening consequences Grade 5: Death related to AE
Number of Serious Adverse Events (SAE) that occurs in Phase 2 | Serious Adverse events will be recorded from informed consent through 28 days (±7 days) after the last dose of study drug
  Results in death, Is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, Is a congenital anomaly or birth defect, Requires intervention to prevent permanent impairment or damage considered as a SAEs
Laboratory Parameters in Phase 2 | For hematology, clinical chemistry and coagulation: at Screening; at Days 1, 8, 15, and 22 of Cycle 1; at Days 1 and 15 of each subsequent treatment cycle (each cycle is 28 days); and at EOT. For urinanalysis: at screening, day 1 of cycle 2 and at EOT
  Incidence of clinically significant clinical laboratory abnormalities (hematology, clinical chemistry, coagulation, and urinalysis)
Vital Signs in Phase 2 | Baseline through study completion, an average of 2 years
  Incidence of clinically significant vital signs abnormalities, including blood pressure, heart rate, respiratory rate, and body temperature.
ECG Parameters in Phase 2 | On Day 1 of cycle 1, 2, 3 and 4. (Each cycle is 28 days)
  Incidence of clinically significant 12-lead ECG abnormalities, assessed from triplicate ECG recordings, including QT/QTc interval.
Chest X-ray (CXR) Abnormalities in Phase 2 | Baseline (Screening) and through study completion, an average of 2 years
  Incidence of clinically significant chest X-ray abnormalities.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF